CLINICAL TRIAL: NCT01353027
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AVI-6002 in Healthy Adult Volunteers
Brief Title: Safety Study of Single Administration Post-Exposure Prophylaxis Treatment for Ebola Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6002-us-101
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Ebola Hemorrhagic Fever
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AVI-6002 (Experimental): Phosphorodiamidate morpholino antisense oligomer with positive charges on selected subunits (PMOplus™)
  Interventions: Drug: AVI-6002

INTERVENTIONS:
Drug: Placebo — Normal saline
  Arms: Placebo
Drug: AVI-6002 — Single intravenous administration
  Arms: AVI-6002

SUMMARY:
The purpose of this study is to characterize the safety and pharmacology of single administrations of AVI-6002, a post-exposure prophylaxis candidate treatment for Ebolavirus.

DETAILED DESCRIPTION:
Ebola hemorrhagic fever (EHF) is a rare human disease caused by Ebola Virus (EBOV), a filamentous single-stranded, negative-sense RNA virus. Since 1976 several Ebolavirus outbreaks have occurred with fatality rates ranging from 57% to 90%, with most of these outbreaks traced to single EBOV species; EBOV-Z. No effective therapy is currently available for Ebolavirus.

AVI-6002 is an experimental combination of 2 phosphorodiamidate morpholino antisense oligomers with positive charges on selected subunits (PMOplus™). These oligomers specifically target viral messenger RNA encoding 2 Ebolavirus proteins thought to be important in viral replication and host immune suppression. The present study is designed to characterize the safety, tolerability and pharmacokinetics of escalating single-administration doses of AVI-6002 in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and between the ages of 18 and 50 years in good general health
* Volunteers must be willing to use barrier methods of contraception or be of non-childbearing potential
* Volunteers must be willing to undergo a urine screen for drugs of abuse

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Any clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology or urinalysis
* Positive test for human immunodeficiency virus, hepatitis B or hepatitis C or known history of HIV infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 28 Days
  The frequency and severity of adverse events will be monitored through 28 days post administration.

SECONDARY OUTCOMES:
Drug concentration in plasma | 28 days
Drug concentration in urine | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: William B Smith, MD, Principal Investigator — New Orleans Center for Clinical Research-Knoxville; Alison Heald, MD, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee, United States